CLINICAL TRIAL: NCT05610150
Title: Cephalometric Changes in Pharyngeal Airway Dimensions After Functional Treatment With Twinblock Versus Myobrace Appliances in Developing Skeletal Class II Patients: A Randomized Clinical Trial
Brief Title: Pharyngeal Airway Dimensions With Twinblock Versus Myobrace Appliances in Developing Skeletal Class II Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0418-03/2022
Record Dates: First submitted 2022-11-02; First posted 2022-11-09 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2022-10

CONDITIONS: Malocclusion, Angle Class II, Division 1
Keywords: Airway; Myobrace; Twinblock
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myobrace functional Appliance (Active Comparator): Thirteen patients with developing skeletal Class II malocclusion will be treated with Myobrace functional appliance for six months.
  Interventions: Device: Myobrace Functional Appliance
- Twin Block Functional appliance (Active Comparator): Thirteen patients with developing skeletal Class II malocclusion will be treated with Twinblock functional appliance for six months.
  Interventions: Device: Twin Block

INTERVENTIONS:
Device: Myobrace Functional Appliance — An Appliance for treating growing Class II patients with mandibular deficiency
  Arms: Myobrace functional Appliance
Device: Twin Block — An Appliance for treating growing Class II patients with mandibular deficiency
  Arms: Twin Block Functional appliance

SUMMARY:
The goal of this clinical trial is to compare the pharyngeal airway changes after treatment with Myobrace and after treatment with Twinblock in developing skeletal Class II patients.

The main question it aims to answer is: Is the efficacy of the twin-block Vs Myobrace appliances in the improvement of pharyngeal airway dimensions in adolescents having skeletal Class II malocclusion with retrognathic mandible utilizing sagittal pharyngeal airway area measurements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children
* 9-12 Years
* Skeletal Class II with mandibular defeciency and normal maxillary growth depending on clinical diagnosis and confirmed with lateral cephalometric x-reay readings ( ANB angle >4 and SNA angle <78)

Exclusion Criteria:

* Previous Orthodontic treatment
* Previous extractions
* mandibular shifts
* Severe Crowding
* Anterior open bite
* Any perioral habits

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
SNA | Six months
  Angle formed between points Sella, Nasion and A point and describes anteroposterior position of the maxilla relative to the anterior cranial base.
SNB | Six months
  Angle formed between points Sella, Nasion and B point and describes anteroposterior position of the mandible relative to the anterior cranial base.
ANB | Six months
  Angle formed between points A, Nasion and B point indicating the skeletal relationship between the maxilla and the mandible.
Witts appraisal | Six months
  The linear distance between the perpendicular projections of points A and B over the functional occlusal plane.
FMA | Six months
  Angle formed between mandibular plane and Frankfort horizontal plane.
Pharyngeal air way area measurement | Six months
  The upper border of Naso Pharyngeal air way area will be delineated by a line extending from the harmonium (H) to the posterior nasal spine. The lower extent of the NPAA will be traced by marking a line at the tip of the soft palate parallel to the Frankfort horizontal (FH) plane extending to the posterior wall of the pharynx. The OPAA and LPAA are differentiated by a line drawn at the level of the tip of epiglottis parallel to the FH plane to the posterior wall of the pharynx. The lower border of the LPAA is defined as a line drawn parallel to FH plane and passing through the anteroinferior most point (C5AI) of the fifth cervical vertebra. Area will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Median, PhD, Study Director — Alexandria University
Locations (1):
- Ahmed Median, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No